CLINICAL TRIAL: NCT02855957
Title: Evaluation of the Free α-hemoglobin Pool in the Red Blood Cells : Prognostic Marker and Severity Index in Thalassemic Syndromes
Acronym: ALPHAPOOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Paris 12 Val de Marne University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P120205
Record Dates: First submitted 2016-07-31; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-07

CONDITIONS: Thalassemic Syndromes
Keywords: Alpha-Hemoglobin Stabilizing Protein; alpha-Hb pool; thalassemias; diagnostic method; biomarker
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood sample (Other): A blood collection is carry out in the three populations of patients during the day of their enrolment.
  Interventions: Other: Free α-Hb pool analysis

INTERVENTIONS:
Other: Free α-Hb pool analysis

SUMMARY:
Our project aims to assess and validate an innovative prognostic and diagnostic test in order to i) define a severity index of the β-thalassemia according to the free α-Hb pool for a better management of the patient; ii) differentiate the α-thalassemia and β-thalassemia and iii) follow the evolution of this pool in response to treatment of patients. In the future, this prognostic test based on the measurement of free α-Hb pool may be suitable for routine laboratory practice. To carry out this project, cohort of 85 thalassemic patients and a group of 50 healthy volunteers have been recruited.

ELIGIBILITY:
Inclusion Criteria Patient

* Age ≥ 18 years
* Written informed consent
* Affiliation to social security
* Known Hb Phenotypes
* Biological phenotype corresponding to a classical picture of thalassemia

Healthy volunteers

* Age ≥ 18 years
* Written informed consent
* Affiliation to social security

Exclusion Criteria Patient

* Transfusion for less than 3 months
* Chronic active viral disease: hepatitis B, C, HIV
* Ongoing infections or known inflammatory diseases
* Hyper or Hypothyroidism known or subject treated by Levothyrox
* Active pathology or tumor remission for less than 5 years
* Oral corticosteroid
* Hemoglobinopathy other than thalassemia for patients
* Treatment by Hydroxyurea for more than 3 months
* Treatment by stimulating agent erythropoiesis for longer than 3 months

Healthy volunteers

* Transfusion for less than 3 months
* Chronic active viral disease: hepatitis B, C, HIV
* Ongoing infections or known inflammatory diseases
* Hyper or Hypothyroidism known or subject treated by Levothyrox
* Active pathology or tumor remission for less than 5 years
* Oral corticosteroid
* Genetically related to person with hemoglobinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Correlation between the pool of free α-Hb and genotype α and β -globin of the patient and if necessary with the genotype AHSP gene | Day 1

SECONDARY OUTCOMES:
Correlation between the pool of free α-Hb and Hb value | Day 1
Correlation between the pool of free α-Hb and Mean Corpuscular Hb | Day 1
Correlation between the pool of free α-Hb and Mean Cell Volume | Day 1
Correlation between the pool of free α-Hb and percent of reticulocytes | Day 1
Correlation between the pool of free α-Hb and fetal Hb | Day 1
Correlation between the pool of free α-Hb and erythrocyte enzymes | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Galacteros, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Vasseur C, Pissard S, Domingues-Hamdi E, Marden MC, Galacteros F, Baudin-Creuza V. Evaluation of the free alpha-hemoglobin pool in red blood cells: a new test providing a scale of beta-thalassemia severity. Am J Hematol. 2011 Feb;86(2):199-202. doi: 10.1002/ajh.21918. PMID 21264907